CLINICAL TRIAL: NCT01685762
Title: Metformin for the Treatment of Endometrial Hyperplasia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1205
Record Dates: First submitted 2012-07-26; First posted 2012-09-14 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2019-01

CONDITIONS: Endometrial Hyperplasia; Endometrial Hyperplasia Without Atypia
Keywords: Endometrial hyperplasia; Uterus; Pilot; Metformin
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin once daily for 4 weeks (weeks 1-4) and then twice daily for 8 weeks (weeks 5-12).
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850 mg of metformin taken once daily by mouth for 4 weeks (weeks 1-4) and then twice daily by mouth for 8 weeks (weeks 5-12).
  Other Names: Fortamet; Glucophage; Glumetza; Riomet

SUMMARY:
The purpose of this study is to see if metformin will be effective in making endometrial hyperplasia without atypia better by returning the tissue to a normal state.

DETAILED DESCRIPTION:
This is a multi-institutional pilot clinical trial designed to estimate the response rate and safety of metformin for the treatment of simple and complex endometrial hyperplasia (EH) without atypia. Enrollment of patients will occur at UNC-Chapel Hill and Southern Pines Women's Health Center. Fifteen patients will be enrolled over the course of 1 year. Metformin will be initiated at 850 mg orally once daily, and titrated up to twice daily over a minimum of 1 months time. Treatment will last 12 weeks and then patients will undergo repeat endometrial biopsy to assess for regression or persistence of EH.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-75 years old
* Have a confirmed diagnosis of endometrial hyperplasia without atypia based upon endometrial biopsy
* Have no contraindications to short-term metformin therapy
* Have a creatinine clearance of ≥ 90 ml/min, as calculated by the Cockroft-Gault formula
* Have normal serum transaminase values (AST and ALT)
* Need to be able to undergo metformin treatment for a duration of 12 weeks prior to repeat endometrial biopsy

Exclusion Criteria:

* Are currently taking metformin or have taken metformin in the past 6 months or have a history of an allergic reaction or intolerance at any time to metformin
* Have a history of liver or renal dysfunction.
* Have a random glucose of ≤ 65 or ≥ 200
* Have a recent history of alcoholism. Former alcoholics who have abstained from alcohol for 5 years or more may be enrolled in this study.
* Have a history of vitamin B12 deficiency
* Are pregnant
* Are currently taking insulin
* Are taking a drug that may significantly interact or influence the metabolism of metformin
* In the opinion of the investigator, the patient is felt not to be appropriate for the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Response Rate | 12 weeks
  Evaluation of hyperplasia resolution by comparison of pre- and post-treatment endometrial biopsies.

SECONDARY OUTCOMES:
Toxicity evaluation | 12 weeks
  Number of subjects who experience side effects
Patient Compliance | 12 weeks
  Percentage of patients successfully completing metformin therapy.
Potential molecular markers in response to treatment with Metformin | 12 weeks
  Compare changes in potential biomarkers, including metabolic factors and molecular markers of downstream targets of the metformin/mTOR signaling pathway, before and after metformin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Southern Pines Women's Health Center, Southern Pines, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org